CLINICAL TRIAL: NCT05678179
Title: Randomized Pilot Study Investigating the Feasibility and Acceptability of Utilizing Telehealth for Increasing Access to Bariatric Surgery
Brief Title: The Feasibility and Acceptability of Utilizing Telehealth for Increasing Access to Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gretchen E. Ames, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-011275
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Telehealth; Face-2-Face (F2F)
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Patients seeking bariatric surgery will be randomized to a Telehealth Treatment Group or a Face-to-Face (F2F) treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental)
  Interventions: Behavioral: Telehealth
- In Person (Face-2-Face) (Active Comparator)
  Interventions: Behavioral: In Person (Face-2-Face)

INTERVENTIONS:
Behavioral: Telehealth — Patients will participate in standard clinical practice for bariatric surgery preparation with 50% of visits occurring via telehealth.
  Arms: Telehealth
Behavioral: In Person (Face-2-Face) — Patients will participate in standard clinical practice for bariatric surgery preparation with face-2-face clinic visits.
  Arms: In Person (Face-2-Face)

SUMMARY:
Bariatric surgery is recommended as the most efficacious treatment for patients living with obesity (body mass index [BMI; kg/m2] > 40; or BMI 35-39.9 with related medical conditions). Adoption of telehealth services offers an opportunity to reduce barriers and expand access to high quality specialty care for patients considering bariatric surgery for treatment of obesity. Two important advances in telehealth services occurred during the COVID-19 public health emergency. Specifically, the patient's home is now the origin site for all services where patients are no longer required to travel to a designated telehealth location, and the use of telehealth has expanded to multidisciplinary health care teams. Our bariatric surgery care team has gained valuable experience using a combination of face-to-face (F2F) and telehealth visits for multidisciplinary evaluation in preparation for bariatric surgery since March 2020. Appointments that do not require a physical exam like nutrition, psychology, group education, and medical visits after completion of pre-operative testing are particularly amenable to telehealth services. Increased use of telehealth has the potential to reduce barriers to care (e.g., lack of access to accredited bariatric surgery treatment centers, extended travel time for multiple pre-surgery appointments), increase adherence to required program visits, and increase patient satisfaction. Patient satisfaction variables may include reduced time away from work, flexibility in appointment scheduling, and reduced physical demands of multiple F2F visits. A necessary first step is to demonstrate that the protocol outlined below can be successfully implemented in a real-world clinical setting and is deemed acceptable by patients preparing for bariatric surgery.

DETAILED DESCRIPTION:
Goals and Objectives

Study participants will be randomized to either a Telehealth treatment group where greater than 50% of visits are conducted via telehealth and testing is completed where the patient resides or to a F2F treatment group. Outcomes will include feasibility and patient acceptability of telehealth visits, adherence to required program visits, program retention, time to surgery, surgery completion, and payment parity data.

Specific aim 1 (primary): The primary aim is to assess the feasibility and acceptability of telehealth for increasing access to bariatric surgery and compare outcomes to patients who receive F2F visits. Feasibility and acceptability were selected as the primary outcomes for this pilot trial because the efficacy of any program is contingent on its ability to be implemented by providers and its acceptability to patients. Hypothesis: The Telehealth treatment group (> 50% of pre-surgery visits telehealth and testing performed locally) will be feasible to implement as evidenced by our ability to recruit and retain participants and acceptable to participants as evidenced by self-report of satisfaction with the program, adherence to required visits, program retention, time to surgery, and completion of surgery. We hypothesize that when comparing the Telehealth and F2F treatment groups, there will be no clinically meaningful differences regarding outcome variables.

Specific aim 2 (secondary): A secondary aim is to compare payment parity between Telehealth and F2F treatment groups. Hypothesis: Telehealth and F2F visits will be similarly reimbursed for bariatric visits.

Study Participants:

Participants will be 50 patients referred for bariatric surgery and who meet medical necessity criteria for bariatric surgery. Potential participants will be contacted regarding participation in the study prior to their first scheduled appointments. Should a patient wish to volunteer for the study, the study coordinator will conduct the screening interview to determine eligibility based on inclusion criteria and review the study protocol. Potential participants will be given the opportunity to ask questions and then will be asked to provide written informed consent. The consent form will clearly explain that participation in the study is voluntary and will not affect current or future care at any Mayo Clinic.

Inclusion Criteria (1) Meet medical necessity criteria for primary bariatric surgery and reside in FL, (2) can participate fully in all aspects of the protocol and keep scheduled appointments, (3) have in home access to telehealth (4) provide written informed consent, (5) are willing to accept randomization, and (6) have a primary care doctor to facilitate local testing in preparation for bariatric surgery.

Procedures and Measures:

This study will employ an unblinded randomized parallel group design. Participants will be randomly assigned to the Telehealth treatment group (N= 25) or the F2F treatment group (N= 25), where the randomization schedule will be determined by the statistician. The protocol is designed to approximate real-world conditions which will enhance generalizability for expansion to all patients who desire bariatric surgery. Permission to collect basic demographic and medical information from participants who decline to participate in the study will be requested. This information will be used to compare the characteristics of individuals who agree to participate in the study versus those who decline participation. Individuals who discontinue study participation any time prior to having bariatric surgery will be contacted to obtain information regarding the reason for discontinuation.

Recruitment:

Patients will be identified consecutively on bariatric medical provider's calendar. The study coordinator will contact those who meet inclusion criteria by phone. If patients agree to participation in the study, oral consent will be obtained. The HIPPA disclosure form will be sent via email to the participant. Participants will return the signed form via email to the study the coordinator.

Outcome Measures:

Telehealth feasibility will be measured by whether >50% of telehealth group visits are conducted virtually, and testing is performed locally. Patients who have complex medical problems may require F2F medical and surgeon visits to be determined by medical and surgical providers.

Patient acceptability will be measured by a questionnaire constructed by the authors to capture the acceptability of participation in the Telehealth treatment group compared to the F2F condition. Responses to Likert scale (5-points) items will be summarized as the mean of all items. The treatment will be considered acceptable if greater than 50% of participants rate satisfaction with a mean score of 4 or greater (e.g., strongly disagree to strongly agree). The survey will be administered to all participants via email using Qualtics.

Program Adherence: Adherence will be measured by whether the patient completed of all visits required for bariatric surgery preparation. No show and reschedule data will be collected from the patient records.

Time to Surgery: The number of days will be from the date of the initial consultation to time of surgery will be counted to determine time to surgery.

Program retention and surgery completion will be compared across groups.

Insurance payer parity will be compared across groups.

Benefits:

Telehealth could potentially expand access to high quality specialty bariatric surgery care for patients living with obesity. This may include patients across Florida (and potentially Georgia with licensure strategy recommendations from the Center for Digital Health) who live in rural and/or underserved communities without access to accredited bariatric surgery programs. All bariatric surgery program licensed providers have been utilizing telehealth technology since March 2020, and these visits are now part of routine care. The bariatric surgery program could potentially be marketed as offering equally efficacious pathways to surgery including F2F or a hybrid schedule of telehealth and F2F visits. With positive results these, pathways could be extended to follow-up care (1, 3, 6, 12-months) in the first year after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

Meet medical necessity criteria for primary bariatric surgery and reside in FL, (2) can participate fully in all aspects of the protocol and keep scheduled appointments, (3) have in home access to telehealth (4) provide written informed consent, (5) are willing to accept randomization, and (6) have a primary care doctor to facilitate local testing in preparation for bariatric surgery.

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Telehealth Feasibility | Pre-surgery
  Telehealth feasibility will be measured by whether >50% of telehealth group visits are conducted virtually, and testing is performed locally.
Telehealth Acceptability | After each provider visit pre-surgery
  Acceptability will be measured by a questionnaire constructed by the authors to capture the acceptability of participation in the Telehealth treatment group compared to the F2F condition. Responses to Likert scale (9-points) items will be summarized as the mean of all items. The treatment will be considered acceptable if greater than 50% of participants rate satisfaction with a mean score of 6 or greater (e.g., satisfied to extremely satisfied). The survey will be administered to all participants via email using Qualtics.

SECONDARY OUTCOMES:
Program Adherence | After each provider visit pre-surgery
  Adherence will be measured by whether the patient completed of all visits required for bariatric surgery preparation. No show and reschedule data will be collected from the patient records.
Time to Surgery | Measured date of surgery.
  Time to surgery will be measured in days from the date of the initial consultation.
Program Retention and Surgery Completion | Pre-surgery
  Retention will be measured by whether the patient completed of all visits required for bariatric surgery preparation. No show and reschedule data will be collected from the patient records. Completion of surgery will be documented.
Insurance Payer Parity | Pre-surgery
  Reimbursement of provider services across groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials